CLINICAL TRIAL: NCT01604161
Title: A Multicentre, Open Label, Non-interventional Study to Evaluate on Long-term Safety and Efficacy of Norditropin® Formulation in Child Patients With GHD or Turner Short Stature Without Closure of Epiphyseal Discs.
Brief Title: Non-interventional Study of Patients Using Norditropin® for Growth Hormone Deficiency or Turner Syndrome
Acronym: NordiPAD
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GH-3910
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Growth Hormone Disorder; Growth Hormone Deficiency in Children; Genetic Disorder; Turner Syndrome
MeSH Terms: conditions — Genetic Diseases, Inborn; Turner Syndrome | interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Somatropin
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — Collection of safety and efficacy data in connection with use of somatropin (Norditropin®) in daily clinical practice.

SUMMARY:
This study is conducted in Japan. The aim of this study is to collect information about the efficacy and safety of Norditropin® (somatropin) in the long-term treatment of short stature with GHD (Growth Hormone Deficiency) where epiphysial discs are not closed and short stature with Turner Syndrome where epiphysial discs are not closed.

ELIGIBILITY:
Inclusion Criteria:

* Growth hormone deficiency or short stature due to Turner Syndrome where the epiphyseal discs are not closed

Exclusion Criteria:

* Diabetic
* Patients with malignant tumors
* Women who are either pregnant or likely to be pregnant
* Known or suspected allergy to study product(s) or related products

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from normal practice who have been deemed appropriate to receive somatropin ( Norditropin®) as part of routine out-patient care by the prescribing physician.
Sampling Method: Non-Probability Sample
Enrollment: 2016 (Actual)
Dates: Start 2005-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in height | Week 0, Month 36, final height is reached
Incidence of adverse reactions (ADRs) | 36 months, accumulation of study period

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com